CLINICAL TRIAL: NCT03445910
Title: Effect of Intrauterine Injection of Human Chorionic Gonadotropin Before Embryo Transfer on Implantation and Pregnancy Rates in Intracytoplasmic Sperm Injection: a Prospective Randomized Study
Brief Title: Intrauterine Injection of Human Chorionic Gonadotrophin and Pregnancy Rate in ICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hayam Fathy Mohammad, Assisted professor of obstetrics and gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2018-02-21; First posted 2018-02-26 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Repeated Implantation Failure
Keywords: human chorionic gonadotropin
MeSH Terms: interventions — Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Investigator
Masking Description: one hundred opaque envelopes will be numbered serially and in each envelope the corresponding letter which denotes the allocated group will be put according to randomization table. Then all envelopes will be closed and put in one box. When the first patient arrives, the first envelope will be opened and the patient will be allocated according to the letter inside.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human chorionic gonadotrophin (Experimental): The hCG Group included 50 patients who had an intrauterine injected of 500 IU of hCG on the day of ovum pick-up
  Interventions: Drug: Human chorionic gonadotropin
- control (No Intervention): The Control Group included 50 patients who went through the ICSI conventional protocol without intrauterine injection.

INTERVENTIONS:
Drug: Human chorionic gonadotropin — intrauterine injected of 500 IU of hCG on the day of ovum pick-up and
  Other Names: Chorimone; pregnyl
  Arms: Human chorionic gonadotrophin

SUMMARY:
Despite recent advances in clinical and laboratory techniques of Assisted Reproductive Technology (ART), the pregnancy rate remains around 30% per cycle. It has been estimated that 50% to 75% of lost pregnancies are due to failure of implantation.

The process of implantation is a locally controlled paracrine/juxtacrine-mediated phenomenon. Successful implantation depends on the synchronized "cross-talk" between a functional blastocyst and a "receptive" endometrium. This process leads to apposition, attachment and invasion of embryos and subsequent normal placentation. So the objective of this study is investigate the impact of intrauterine injection of human chorionic gonadotropin (hCG) at the day of ovum pick-up on implantation and pregnancy rates in patients with recurrent implantation failure.

DETAILED DESCRIPTION:
The endometrium can only support implantation during a discrete period of about 6 to 9 days after LH peak; termed the "window of implantation". During this period endometrial glandular epithelium is differentiated into a highly secretory state with the production of various cytokines and growth factors that facilitate implantation. In fact, several substances secreted from the embryo or the endometrium affect implantation. These include cyclic adenosine monophosphate, relaxin, gonadotropin, prostaglandin E2, and glycoprotein hormones.

Human chorionic gonadotropin (hCG) is the earliest blastocyst-derived signals received by the endometrium; it is transcribed as early as the 2-cell embryo stage. It is produced by the trophectodermal cells of the preimplantation blastocyst. Recent evidence suggests that hCG is also produced by the endometrial epithelial cells during the secretory.

It has been shown that intrauterine injection of hCG before embryo transfer significantly improves pregnancy rates in IVF/ICSI cycles.

ELIGIBILITY:
Inclusion Criteria:

A- Age between 20 and 35 years old.

B- Patients undergoing ICSI trial after one or more previous failure.

Exclusion Criteria:

A- Females with any local cause, uterine pathology, e.g: uterine myoma or previous myomectomy, endometriosis or the presence of hydrosalpinges.

B- Patients undergoing ICSI trial for the first time.

C- Previous Asherman Syndrome.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
implantation rate | six weeks from the last menstrual period
  is defined as the number of gestational sacs observed at echographic screening at 6 weeks of pregnancy divided by the number of embryos transferred

SECONDARY OUTCOMES:
biochemical pregnancy | two weeks following embryo transfere
  defined as positive from quantitative values of serum test of β human chorionic gonadotropin according to standard values that are used in the laboratory.
clinical pregnancy | eight weeks from last menstrual period
  is defined as viable pregnancy when there is evidence of gestational sac, embryo and fetal heart activity at time of trans-vaginal ultrasound evaluation by the 8th week.

CONTACTS AND LOCATIONS:
Overall Officials: Hayam F Mohammad, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No